CLINICAL TRIAL: NCT03711409
Title: Comparison of Soft Tissue Biased Manual Therapy and Conventional Physical Therapy on Shoulder Kinematics, Muscle Performance, Functional Impairment & Pain in Patients With Frozen Shoulder
Brief Title: Comparison of Soft Tissue Biased Manual Therapy and Conventional Physical Therapy in Patients With Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, Department of Physical Therapy and Assistive Technology, National Yang-Ming University, National Yang Ming Chiao Tung University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCHIRB-10705119-E
Record Dates: First submitted 2018-08-06; First posted 2018-10-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Frozen Shoulder; Shoulder Adhesive Capsulitis
Keywords: Frozen Shoulder; Manual therapy; Soft tissue mobilization
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Subjects are divided into soft tissue biased manual therapy group and conventional physical therapy group by two different hospitals
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft tissue biased manual therapy group (Experimental): It includes hot pack and muscle release technique of the muscles around the shoulder. The patient receives treatment 45 minutes per times and 2 times per week for 6 weeks.
  Interventions: Other: Soft tissue biased manual therapy group
- Conventional physical therapy group (Experimental): It includes modality (electrotherapy, ultrasound and low-level laser therapy) and GH joint mobilization. The patient receives treatment 45 minutes per times and 2 times per week for 6 weeks.
  Interventions: Other: Conventional physical therapy group

INTERVENTIONS:
Other: Soft tissue biased manual therapy group — It includes hot pack and muscle release technique of pectoralis major, pectoralis minor, teres major, teres minor, infraspinatus and posterior deltoid muscles. Subjects are supine on the bed. The muscle release technique is applied at the end available range and the acceptable intensity. The time of muscle release intervention is about 30 min and hot-pack about 15 min.
  Arms: Soft tissue biased manual therapy group
Other: Conventional physical therapy group — It includes modality (electrotherapy, ultrasound and low-level laser therapy) and GH joint mobilization. GH joint mobilization includes anterior to posterior glide, caudal glide and distraction. The intensity of joint mobilization is grade III to IV. The time of joint mobilization is about 30 min and hot-pack for 15 min.
  Arms: Conventional physical therapy group

SUMMARY:
Adhesive capsulitis, also known as frozen shoulder (FS), is a condition characterized by the functional restriction of both active and passive shoulder motion with unremarkable glenohumeral joint radiographs findings. Shoulder pain almost exists during the whole course of frozen shoulder. Pain induces muscle spasm and causes pain-spasm-pain cycle resulting in limited range of motion, changed muscle recruitment pattern and finally influences neuromuscular control. Commonly used conservative interventions for FS patients include joint mobilization, corticosteroid injection, exercise, modality and soft tissue mobilization. Despite joint mobilization is the most commonly used manual therapy in patients with FS, the evidence level is weak and the efficacy is not superior to other conservative treatments. Soft tissue mobilization is widely used in lots of musculoskeletal conditions. The effects of soft tissue mobilization include breaking the adhesion tissue and improving range of motion, muscle strength and motor control. However, few studies have investigated the effect of soft tissue mobilization in patients with frozen shoulder. Therefore, the purpose of this study is to investigate and compare the effect of soft tissue biased manual therapy and conventional physical therapy in patients with primary FS.

DETAILED DESCRIPTION:
Adhesive capsulitis, also known as frozen shoulder (FS), is a condition characterized by a functional restriction of both active and passive shoulder motion with unremarkable glenohumeral joint radiographs findings. Frozen shoulder is divided into primary and secondary type. The mechanism of primary FS is still unknown and the secondary FS may accompany with shoulder injuries. The incidence of primary FS is 2 to 5.8% and the risk factors are diabetes and thyroid disease.

The course of FS is divided into four consecutive stages which are inflammation, painful, frozen and thawing phase. Shoulder pain almost exists during the whole course of frozen shoulder. The pain and discomfort of FS patients are frequently localized to the deltoid insertion and coracoid process. Pain induces muscle spasm and causes pain-spasm-pain cycle resulting in limited range of motion, changed muscle recruitment pattern and finally influences neuromuscular control.

Commonly used conservative interventions for FS patients include joint mobilization, corticosteroid injection, exercise, modality and soft tissue mobilization. Despite joint mobilization is the most commonly used manual therapy in patients with FS, the evidence level is weak and the efficacy is not superior to other conservative treatment s. Soft tissue mobilization is widely used in lots of musculoskeletal conditions. The effects of soft tissue mobilization include breaking the adhesion tissue and improving range of motion, muscle strength and motor control. However, few studies have investigated the effect of soft tissue mobilization in patients with frozen shoulder. Only one study used one-time muscle release to FS patients and investigate improvement in shoulder biomechanics, muscle strength and ROM. Therefore, the purpose of this study is to investigate and compare the effect of soft tissue biased manual therapy and conventional physical therapy for six weeks in patients with primary FS.

The study design is a pretest-posttest control group design. The investigators plan to recruit 70 patients with primary frozen shoulder and divide them into a soft tissue biased manual therapy group and a conventional physical therapy group. The sample size is determined by the previous study. It is based on a significance level of 0.05, and a power of 0.80. The outcome measures in this study include scapula kinematics, scapula position, the range of motion, muscle tone, muscle strength, pain and functional impairment.

LIBERTY™ electromagnetic tracking system (Polhemus, Colchester, VT, USA) was used to collect three-dimensional kinematic (3D) data during scaption, hand to neck and hand to back tasks at a sampling rate of 120 Hz, and the software Motion Monitor® (Innovative Sport Training, Inc., Chicago. IL. USA) was used to analyze the data. The main measurements of shoulder kinematics include scapular upward/downward rotation, internal/external rotation, and anterior/posterior tilt. A stylus was used to digitize the bony landmarks for defining the anatomical coordinate system. The methods for this measure have been described previously.

For collecting muscle activation data, the investigators used surface electromyography (sEMG, TeleMyo 2400 G2 Telemetry; Noraxon USA, Inc., USA) to collect scapular muscles' activation during those tasks. The investigators will measure the muscle activities of the pectoralis major, upper trapezius, infraspinatus, teres major and lower trapezius. The electrodes will be placed according to previous studies and be positioned in parallel to the direction of the muscle ﬁbers.

The range of motion of shoulder flexion, abduction, external rotation and internal rotation will be measured by plastic universal goniometer according to Norkin's methods. The muscle strength of lower trapezius, external rotators and internal rotators are measured by the hand-held dynamometer. The scapula positions are measured by modified scapular sliding test with calliper during arms by sides, hands on the hips and scaption 90 degrees. The muscle tone of pectoralis major, upper trapezius, infraspinatus and teres complex will be measured by hand-held myotonometer (Myoton-Pro, Myoton AS, Tallinn, Estonia) in shoulder resting position according to previous studies. The functional impairments are measured by Flexilevel Scale of Shoulder Function questionnaire. The pain level is measured by the visual analogue scale.

Participants in the soft tissue biased manual therapy group will receive heat and muscle release for six weeks and participants in conventional physical therapy group will receive modalities and joint mobilization for six weeks. The measurement will be obtained at baseline, 3 weeks, and after the intervention. Repeated measures ANOVA will be used for data analysis. The level of significance sets at α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Primary adhesive capsulitis diagnosed by orthopaedic surgeon or physiatrist
* Reduction in range of motion in more than two planes
* < 30 degrees of the external rotation range of motion during shoulder abduct to 90 degree
* No radiologic abnormality
* Onset time more than three months
* No night pain and resting pain

Exclusion Criteria:

* History of stroke, diabetes mellitus, rheumatoid arthritis, rotator cuff tear, shoulder osteoarthritis, surgical stabilization/surgery of the shoulder, osteoporosis, or malignancies in the shoulder region

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Scapulo-humeral rhythm (scapular kinematics) during functional movements | Baseline and after 6-week intervention
  Change from baseline of scapular kinematics to after 6 week intervention during scaption task, hand to neck task and hand to back task

SECONDARY OUTCOMES:
Range of motion of shoulder joint (Goniometer) | Baseline, 3-week intervention and 6-week intervention
  Shoulder range of motion in degree of flexion, abduction, internal rotation and external rotation
Mechanical stress relaxation time (ms) of shoulder muscles | Baseline, 3-week intervention and 6-week intervention
  We use Myotometer to measure mechanical stress relaxation time (ms) of pectoralis major, infraspinatus, teres complex and upper trapezius
Creep of shoulder muscles | Baseline, 3-week intervention and 6-week intervention
  We use Myotometer to measure creep of pectoralis major, infraspinatus, teres complex and upper trapezius
Oscillation frequency (Hz) of shoulder muscles | Baseline, 3-week intervention and 6-week intervention
  We use Myotometer to measure oscillation frequency (Hz) of pectoralis major, infraspinatus, teres complex and upper trapezius
Dynamic stiffness (N/m) of shoulder muscles | Baseline, 3-week intervention and 6-week intervention
  We use Myotometer to measure dynamic stiffness (N/m) of pectoralis major, infraspinatus, teres complex and upper trapezius
Muscle strength of shoulder muscles (Hand-held Dyanometer) | Baseline, 3-week intervention and 6-week intervention
  Shoulder muscle strength in Kgw of lower trapezius, internal rotators and external rotators
Scapula dyskinesia | Baseline, 3-week intervention and 6-week intervention
  Use modified lateral scapular slide test to measure during arms by sides, hands on hips and scaption movement
Shoulder disability | Baseline, 3-week intervention and 6-week intervention
  Use Flexilevel Scale of Shoulder Function (Flex-SF) questionnaire Chinese version to measure the disability level of frozen shoulder patients. Flex-SF uses 4-point Likert Scale to measure the disability level. Subjects need to answer a routing question and subgroup them into three different difficulty level. The scores range from 1 to 48 (1= most disable, 48= least disable).
Shoulder pain | Baseline, 3-week intervention and 6-week intervention
  Use visual analogue scale to measure shoulder pain of frozen shoulder patients. We will provide subjects a 10-cm scale for them to point the intensity of their pain (on a 10-cm scale, 0 cm = no pain, 10 cm = the most severe pain).
Scapula motor control (muscle activation percentage) | Baseline and after 6-week intervention
  Change from baseline of scapular muscles' activation in percentage during scaption, hand to neck and hand to back task to after 6-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shih Yi-Fen, PhD, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming University
Locations (1):
- National Yang Ming University, Taipei, Taiwan